CLINICAL TRIAL: NCT05729477
Title: A Prospective Multicenter Study To Assess The Clinical Outcomes Of Current Phacoemulsification Approach To Cataract Extraction Versus The Micor System Device Using Low Energy Lens Extraction In Patients Undergoing Cataract Surgery
Brief Title: A Prospective Multicenter Study To Assess The Clinical Outcomes Of Current Phacoemulsification Approach To Cataract Extraction Versus The Micor System Device
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MICOR-304-102
Record Dates: First submitted 2022-11-08; First posted 2023-02-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Intervention Model Description: The miCOR System used during cataract surgery is a lens fragmentation and lens removal device which is an alternative to conventional phacoemulsification. The miCOR system has no cavitation and no thermogenic energy in the eye which can eliminate the generation of heat inside the eye while at the same time maintaining the same minimally invasive surgical approach through a small clear-cornea 2.5 mm incision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group 1 Phaco Subject Cohort (Active Comparator): The Group 1 Phaco subject cohort will begin enrolling subjects sequentially in the first initial arm of the study with up to 250 eyes total.
  Interventions: Device: Phaco Subject Cohort
- Group 2 miCOR System Subject Cohort (Active Comparator): The Group 2 MICOR System subject cohort, non-use of miLOOP will enroll subsequently with up to 250 eyes total.
  Interventions: Device: miCOR System
- Group 3 miCOR System Subject Cohort (Active Comparator): The Group 3 MICOR System subject cohort, use of miLOOP optional will enroll subsequently with up to 250 eyes total.
  Interventions: Device: miCOR System

INTERVENTIONS:
Device: miCOR System — The miCOR system is a lens fragmentation device used to break up the cataract prior to IOL implantation during cataract surgery.
  Arms: Group 2 miCOR System Subject Cohort; Group 3 miCOR System Subject Cohort
Device: Phaco Subject Cohort — Phaco Subject Cohort
  Arms: Group 1 Phaco Subject Cohort

SUMMARY:
The purpose of this research study is to evaluate the clinical outcomes of current phacoemulsification approaches to cataract extraction involving high-frequency thermogenic energy versus the use of the MICOR System device using low-energy segment removal with a micro-interventional irrigation/aspiration port to evacuate the lens in subjects undergoing routine cataract surgery.

DETAILED DESCRIPTION:
This is prospective, multicenter, 3-arm study designed to provide longitudinal, observational, clinical outcome data for the use of traditional phacoemulsification for subjects undergoing cataract surgery versus the MICOR System device used to evacuate the lens prior to intraocular lens insertion and cataract surgery. Only FDA cleared phacoemulsification devices can be used per indications.

Both eyes of the study subjects may be enrolled into the study; however, if only 1 eye is eligible for study participation, then the eligible eye of the subject may be enrolled. Up to 750 eyes will be enrolled into one of three study groups, up to 250 subjects per group, with a maximum of 10 study centers. The 3 arms of the study groups are as follows:

* Group 1 Phaco subject cohort.
* Group 2 MICOR System subject cohort, non-use of miLOOP.
* Group 3 MICOR System subject cohort, use of miLOOP optional.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand study requirements, willing to follow study instructions and willing to return for required study follow-up visits.
2. Willing and able to understand and complete the informed consent document.
3. Subjects with a cataract grade of 1 to 4+ and are scheduled to undergo cataract surgery.
4. Subjects ≥ 18 years of age.

Exclusion Criteria:

1. Subjects, who in the opinion of the investigator, have "compromised" eye(s); no comorbidities and no patients undergoing concurrent corneal surgery with cataract extraction.
2. Concurrent participation or participation in any clinical trial up to 30 days prior to preoperative visit.
3. Subjects that are pregnant, lactating or planning to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
UCVA Measurement | 1 day postoperative
  The visual acuity measurement after cataract surgery

OTHER OUTCOMES:
Rate of intraoperative and postoperative adverse events. | All adverse events will be followed for 1 month
  All adverse events will be recorded and followed for safety purposes.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Argus Research at Cape Coral Eye Center, Cape Coral, Florida
  - Mittleman Eye, West Palm Beach, Florida
  - Wolfe Eye Clinic, Hiawatha, Iowa
  - Penn State Health Eye Center, Hershey, Pennsylvania
  - Virginia Eye Consultants, Norfolk, Virginia
  - The eye Centers of Racine and Kenosh, Racine, Wisconsin